CLINICAL TRIAL: NCT00295386
Title: Cognitive-Behavioural and Hypnotic Treatment of Chronic Primary Insomnia Among the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bergen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REK Vest nr. 186.03
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; zopiclone

INTERVENTIONS:
Behavioral: Cognitive behavior therapy (CBT)
Drug: Zopiclone

SUMMARY:
The present study examines the short- and long-term clinical efficacy of cognitive-behavior therapy and pharmacological treatment in patients suffering from late-life primary insomnia. 46 subjects suffering from chronic primary insomnia were randomized into either cognitive-behavior therapy (CBT, n=18), hypnotics (7.5 mg Zopiclone, n=16), or placebo treatment (n=12). All active treatments lasted 6 weeks with follow-ups conducted at 6 months. Ambulant clinical polysomnography (PSG) and sleep diaries were used on all three assessment points.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or older
* fulfilment of the DMS-IV criteria for insomnia, including difficulties initiating sleep, maintaining sleep, and/or early morning awakenings with no ability of return to sleep
* duration of at least 3 months
* complaints of impaired daytime functioning.

Exclusion Criteria:

* use of hypnotic medication the last 4 weeks before project start
* use of antidepressive or antipsychotic medications
* signs of dementia or other serious cognitive impairment defined by a score under 25 on the Mini-Mental State Examination
* presence of a major depressive disorder or other severe mental disorder as identified by a clinical assessment based on The Structured Clinical Interview for DSM-IV (SCID-I)
* presence of sleep apnea defined as (A/H index > 15) or periodic limb movements during sleep (PLM index with arousal > 15),
* working nightshifts and unable or unwilling to discontinue this work pattern,
* willingness or inability to stop taking sleep medication before start
* having a serious somatic conditions preventing further participation

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inger H Nordhus, PhD, Study Director — University of Bergen
Locations (1):
- University of Bergen, Bergen, Bergen, Norway

REFERENCES:
- [Result] Sivertsen B, Omvik S, Pallesen S, Bjorvatn B, Havik OE, Kvale G, Nielsen GH, Nordhus IH. Cognitive behavioral therapy vs zopiclone for treatment of chronic primary insomnia in older adults: a randomized controlled trial. JAMA. 2006 Jun 28;295(24):2851-8. doi: 10.1001/jama.295.24.2851. PMID 16804151
- [Result] Omvik S, Sivertsen B, Pallesen S, Bjorvatn B, Havik OE, Nordhus IH. Daytime functioning in older patients suffering from chronic insomnia: treatment outcome in a randomized controlled trial comparing CBT with Zopiclone. Behav Res Ther. 2008 May;46(5):623-41. doi: 10.1016/j.brat.2008.02.013. PMID 18417099
- [Result] Sivertsen B, Omvik S, Havik OE, Pallesen S, Bjorvatn B, Nielsen GH, Straume S, Nordhus IH. A comparison of actigraphy and polysomnography in older adults treated for chronic primary insomnia. Sleep. 2006 Oct;29(10):1353-8. doi: 10.1093/sleep/29.10.1353. PMID 17068990